CLINICAL TRIAL: NCT06915870
Title: Comparison of Empagliflozin and Dapagliflozin in Patients With Heart Failure Taking Standard Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Maqsood (Other Government)
Responsible Party: Sponsor-Investigator, Fatima Maqsood, Head of the Department of Cardiology, Sheikh Zayed Medical College
Organization: Sheikh Zayed Medical College (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 271
Record Dates: First submitted 2025-03-27; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus; Heart Failure
Keywords: ejection fraction; angiotensin receptor neprilysin inhibitor; Dapagliflozin; Empagliflozin
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure | interventions — dapagliflozin; empagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In group A, patients were prescribed Dapagliflozin 10 mg daily for 12 weeks (Experimental): 108 patients fulfilling the selection criteria were enrolled from OPD. Informed consent and demographic data of all the patients were obtained. Then patients were randomly divided in two groups by using lottery method. In group A, patients were prescribed Dapagliflozin 10 mg daily for 12 weeks
  Interventions: Drug: Dapagliflozin 10 mg daily
- In group B, patients were prescribed Empagliflozin 10 mg daily for 12 weeks (Experimental): In group B, patients were prescribed Empagliflozin 10 mg daily for 12 weeks. Standard SGLT2 and ARNI treatment was given as per standard protocol. All patients were followed-up in OPD after 12 weeks for assessment of ejection fraction by using echocardiography
  Interventions: Drug: Empagliflozin 10 MG OD

INTERVENTIONS:
Drug: Dapagliflozin 10 mg daily — Dapagliflozin 10 mg daily for 12 weeks. Standard SGLT2 and ARNI treatment was given as per standard protocol. All patients were followed-up in OPD after 12 weeks for assessment of ejection fraction by using echocardiography
  Arms: In group A, patients were prescribed Dapagliflozin 10 mg daily for 12 weeks
Drug: Empagliflozin 10 MG OD — Empagliflozin 10 mg daily for 12 weeks. Standard SGLT2 and ARNI treatment was given as per standard protocol. All patients were followed-up in OPD after 12 weeks for assessment of ejection fraction by using echocardiography
  Arms: In group B, patients were prescribed Empagliflozin 10 mg daily for 12 weeks

SUMMARY:
Participants were enrolled and randomly divided in two groups. In group A, participants were prescribed Dapagliflozin 10 mg daily. In group B, participants were prescribed Empagliflozin 10 mg daily. All participants were followed-up in OPD after 12 weeks for assessment of ejection fraction.

DETAILED DESCRIPTION:
This study's rationale is to examine the effects of dapagliflozin and empagliflozin on heart failure in patients receiving ARNI and SGLT2. Research revealed that the two medications results are identical. Although the cardiac functioning improved better with empagliflozin. But limited data has been available in this regard, while no local trial conducted before. Thus, in routine SGLT2 and ARNI are given to control glycemic level and maintain cardiac functioning. However, addition of Empagliflozin and Dapagliflozin can be more beneficial in improving cardiac functioning and reducing adverse events. Therefore the investigators planned to conduct this study to get evidence in local population. This will help to improve practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-60 years of either gender diagnosed with heart failure ( Heart failure was defined as presence of ejection fraction <50% on echocardiography, with pedal edema, water in lungs, paroxysmal nocturnal dyspnea or exertional limitation due to failure of ventricular fillings)
* Diabetic patients, with HBA1c>6.5% for >1 year already taking SGLT-2 and ARNI inhibitor.

Exclusion Criteria:

* Patients already had valvular device, mitral or aortic valve regurgitation or stenosis detected on echocardiography, heart transplantation, chronic renal failure or dialysis patients, cardiomyopathy, liver failure or malignancy.
* Patients already taking trial drugs or other anti-glycemic or cardiac medication.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Comparison of Empagliflozin and Dapagliflozin in heart failure in diabetic patients taking Sodium-glucose cotransporter-2 and angiotensin receptor neprilysin inhibitor | 12 weeks
  Participants fulfilling criteria were included. Baseline ejection fraction was calculated. Total 12 weeks of therapy was given. One group was administered dapagliflozin where as empagliflozin was administered to other group. Any variation in condition was assessed by ejection fraction findings of both groups after 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shaikh Zayed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No